CLINICAL TRIAL: NCT01322230
Title: Randomized Trial of Educational Outcomes of WISE-MD
Brief Title: Trial of Educational Outcomes of WISE-MD
Acronym: WISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Augusta University (Other); University of Nebraska (Other); University of Vermont (Other); New York Medical College (Other); State University of New York - Downstate Medical Center (Other); Jefferson Medical College of Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single
Other Study IDs: 1LM009538-R01
Record Dates: First submitted 2011-03-21; First posted 2011-03-24 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Surgery
Keywords: Instructional Design; Online learning module; Surgical education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Experimental): Screen shots with voiceover and no interactivity
  Interventions: Other: Control
- WISEMD Original (Experimental): Learner control of pacing through multi-media content
  Interventions: Other: WISEMD Original
- Social Networking (Experimental): social networking features (Forum and Social Presence)
  Interventions: Other: Social Networking
- Social Networking plus Emotional Design (Experimental): Social networking features plus user interface enhancements
  Interventions: Other: Social Networking plus Emotional Design

INTERVENTIONS:
Other: Control — Multimedia Control
  Other Names: Multimedia Control
  Arms: Control
Other: WISEMD Original — Current WISEMD
  Arms: WISEMD Original
Other: Social Networking — Social networking feature
  Arms: Social Networking
Other: Social Networking plus Emotional Design — social networking features plus user interface enhancements
  Arms: Social Networking plus Emotional Design

SUMMARY:
The purpose of this study is to compare the educational efficacy of instructional design enhancements in on-line learning modules in the context of clinical medical education.

DETAILED DESCRIPTION:
This study involved medical students from seven US medical schools participating in a trial of two WISE-MD computer-based learning modules. Students were randomized to 1 of 4 study arms. The 4 content-equivalent conditions were: screen shots with voiceover and no interactivity; learner control of pacing through multi-media content; social networking features; and social networking features plus user interface enhancements.

ELIGIBILITY:
Inclusion Criteria:

* All third-year medical students at all of the 7 collaborating schools (N= 2308) rotating through the surgery clerkship from July 2009 and September 2011.

Exclusion Criteria:

* Students who do not consent to participate and who decide to withdraw from participation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1363 (Actual)
Dates: Start 2008-10; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Immediate Post Knowledge Test | Week 2
  An 8 week-long Surgery Clerkship (Jefferson University is 12 weeks) occurs 6 times (JU 4 times) per year. Students enroll on day 1, complete the baseline surveys in week 1, access the intervention modules by week 2. Learning outcomes (knowledge test) are measured immediately after the modules, at week 4 they complete online multiple-choice tests and a clinical reasoning measure, week 8, week 12 at JU, students complete a clinical reasoning measure.
Mid-clerkship Knowledge Test | Week 4
  An 8 week-long Surgery Clerkship (Jefferson University is 12 weeks) occurs 6 times (JU 4 times) per year. Students enroll on day 1, complete the baseline surveys in week 1, access the intervention modules by week 2. Learning outcomes (knowledge test) are measured immediately after the modules, at week 4 they complete online multiple-choice tests and a clinical reasoning measure, week 8, week 12 at JU, students complete a clinical reasoning measure.
Mid-clerkship Clinical Reasoning Test | Week 4
  An 8 week-long Surgery Clerkship (Jefferson University is 12 weeks) occurs 6 times (JU 4 times) per year. Students enroll on day 1, complete the baseline surveys in week 1, access the intervention modules by week 2. Learning outcomes (knowledge test) are measured immediately after the modules, at week 4 they complete online multiple-choice tests and a clinical reasoning measure, week 8, week 12 at JU, students complete a clinical reasoning measure.
End-clerkship Clinical Reasoning Test | Week 8
  An 8 week-long Surgery Clerkship (Jefferson University is 12 weeks) occurs 6 times (JU 4 times) per year. Students enroll on day 1, complete the baseline surveys in week 1, access the intervention modules by week 2. Learning outcomes (knowledge test) are measured immediately after the modules, at week 4 they complete online multiple-choice tests and a clinical reasoning measure, week 8, week 12 at JU, students complete a clinical reasoning measure.

SECONDARY OUTCOMES:
Students Baseline Characteristics | Immediately after consenting to participate - Day 1
  The baseline characteristics measure include measures of self-regulation, surgery specific self-efficacy, surgery specific task values, and goal orientation.

CONTACTS AND LOCATIONS:
Overall Officials: Adina Kalet, M.D., M.P.H., Principal Investigator — NYU Langone Health
Locations (7):
- United States (7):
  - Medical College of Georgia, Augusta, Georgia
  - University of Nebraska Medical Center, Omaha, Nebraska
  - SUNY Downstate Medical Center, Brooklyn, New York
  - New York University School of Medicine, New York, New York
  - New York Medical College, Valhalla, New York
  - Jefferson Medical College, Philadelphia, Pennsylvania
  - University of Vermont, Burlington, Vermont

REFERENCES:
- [Background] Kalet AL, Coady SH, Hopkins MA, Hochberg MS, Riles TS. Preliminary evaluation of the Web Initiative for Surgical Education (WISE-MD). Am J Surg. 2007 Jul;194(1):89-93. doi: 10.1016/j.amjsurg.2006.12.035. PMID 17560916